CLINICAL TRIAL: NCT00456989
Title: Phase I/II Study of Docetaxel (Taxotere) in Combination With Doxorubicin HCI Liposome Injection (Doxil) in Advanced Androgen-Independent Prostate Cancer (AIPC)
Brief Title: Study of Taxotere and Doxil to Treat Advanced Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 575-03
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: Androgen Independent; Prostate Cancer; Taxotere; Doxil; AIPC; Advanced Androgen-Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Taxotere and Doxil (Experimental): Treatment will be repeated every 28 days. Taxotere is administered on days 1, 8 and 15 (rate: 1 hour). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 25 and 30, respectively. Treatment will be administered on an outpatient basis. Treatment will be repeated every 28 days. Doxil is administered on day 1 (rate: 1mg/min). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 30 and 30, respectively.
  Interventions: Drug: Taxotere; Drug: Doxil

INTERVENTIONS:
Drug: Taxotere — Treatment will be administered on an outpatient basis. Treatment will be repeated every 28 days. Taxotere is administered on days 1, 8 and 15 (rate: 1 hour). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 25 and 30, respectively.
Drug: Doxil — Treatment will be administered on an outpatient basis. Treatment will be repeated every 28 days. Doxil is administered on day 1 (rate: 1mg/min). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 30 and 30, respectively.

SUMMARY:
This clinical research study is being done because there is no effective treatment for advanced androgen-independent prostate cancer. This study will determine if the combination of medications (Taxotere and Doxil) are effective in this kind of cancer.

DETAILED DESCRIPTION:
Each cycle of treatment will consist of four weeks. The 2 types of medicines are given intravenously (in a vein). Doxil is given on the first day of each cycle. Taxotere is given once a week for the first 3 weeks of each cycle. This is followed by a week of rest until the next cycle starts. Treatment is given on an outpatient basis and hospitalization is not anticipated.

Prior to entry on this study, "screening" tests are performed to determine eligibility to participate. This will involve a complete history and physical examination, vital signs, pain assessment, blood tests including CBC (complete blood count), serum chemistry, and PSA (prostate specific antigen), x-rays (chest x-ray, possible plain films of bones if there are abnormal findings on bone scan for clarification), computerized tomography (CT) scans of the abdomen and pelvis, bone scans, a MUGA scan or 2-D echocardiogram, and a quality of life questionnaire.

After treatment starts the following tests are done to regularly monitor for beneficial and toxic effect of the treatment:

Every week: blood tests.

Every month: physical examination, weight, vital signs (blood pressure, respiration, temperature and heart rate) and PSA test.

Every 2 months: pain assessment, quality of life questionnaire, x-rays (chest x-ray and possible pain films of bones if positive findings are seen on bone scan), computerized tomography (CT) scans (abdomen and pelvis) and bone scans.

Participants may continue with any procedures that are part of their regular cancer care. It is anticipated that participants will be in the study for a minimum of 2 months and as long as they are benefiting from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate.
* Androgen-independent disease progression, as shown by:
* A castrate testosterone level of < 40 ng/dl (this measurement is required only for patients treated with medical testicular suppression). If testicular suppression is achieved medically, treatment to maintain castrate levels of testosterone must be applied continuously.
* A PSA level of at least 4 ng/ml, and rising (with an absolute change of at least 1 ng/ml) on two consecutive measurements at least 2 weeks apart prior to study entry.
* Patients must be off anti-androgens such as flutamide (Eulexin) or nilutamide (Nilandron) for at least four weeks, and six weeks for bicalutamide (Casodex), without evidence of response; or have evidence of progression since anti-androgen withdrawal.
* None or one previous cytotoxic therapy is allowed. (For this study, a combination of agents given at the same period of time is considered one chemotherapy treatment)
* Age > 18 years of age.
* Life expectancy of greater than 12 weeks.
* ECOG performance status 0, 1 or 2 (Karnofsky >50%; see Appendix B).
* Patients must have adequate bone marrow function as defined below:

  * absolute neutrophil count > 1,500/ul
  * platelets > 100,000/ul
  * hemoglobin > 8 g/dl
* Patients must have adequate liver function as defined below:

  * total bilirubin normal, albumin > 3.0 g/dl, and no ascites
  * AST(SGOT) and ALT(SGPT) and Alkaline Phosphatase must be within the range allowing for eligibility
* Patients must have adequate renal function as defined by a creatinine < 2.5 mg/dl or a creatinine clearance > 30 mL/min (measured or estimated by the Cockroft formula) for patients with creatinine levels above 2.5 mg/dl
* Patients must have recovered from acute toxicities from chemotherapy or radiotherapy administered prior to entering this study. Alopecia may not be resolved and peripheral neuropathy (grade 1) may be present.
* Patients must have a MUGA scan or 2-d echocardiogram indicating an ejection fraction of > 50% within 42 days prior to first dose of study drug. The method used at baseline must be used for later monitoring.
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who have had two or more prior chemotherapy treatment(s) (For this study, a combination of agents given at the same period of time is considered one chemotherapy treatment).
* Patients receiving any other investigational agent(s).
* Patients with symptomatic brain metastases or actively receiving any therapy for brain metastasis (because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events).
* Active second malignancy in the last 5 years except for non-melanoma skin cancer or carcinoma-in-situ.
* History of cardiac disease, with New York Heart Association Class II or greater, or clinical evidence of congestive heart failure.
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL, the components of Doxil, docetaxel or other drugs formulated with polysorbate 80.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damian Laber, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Laber DA, Eatrides J, Jaglal MV, Haider M, Visweshwar N, Patel A. A phase I/II study of docetaxel in combination with pegylated liposomal doxorubicin in metastatic castration-resistant prostate cancer. Med Oncol. 2020 Sep 26;37(10):95. doi: 10.1007/s12032-020-01420-7. PMID 32979106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Taxotere and Doxil
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Taxotere and Doxil
Number analyzed (Participants) | 39
Age, Customized [Number; unit: Participants]
  >=18 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose and Toxicity Profile
Time Frame: 2 years
Population: Study was terminated and PI has left the institution. Sincere efforts were made to gather and report the data, however, no data is available for the study
Arm/Group | Taxotere and Doxil
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate
Description: Data not analyzed, PI left institution
Time Frame: 7 years
Population: There is no data to report. Data for this trial was not analyzed, the PI left institution.
Groups:
- Taxotere and Doxil: There is no data to report. Data for this trial was not analyzed, the PI left institution.
  Treatment will be repeated every 28 days. Taxotere is administered on days 1, 8 and 15 (rate: 1 hour). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 25 and 30, respectively. Treatment will be administered on an outpatient basis. Treatment will be repeated every 28 days. Doxil is administered on day 1 (rate: 1mg/min). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 30 and 30, respectively.
  Taxotere: Treatment will be administered on an outpatient basis. Treatment will be repeated every 28 days. Taxotere is administered on days 1, 8 and 15 (rate: 1 hour). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 25 and 30, respectively.
  Doxil: Treatment will be administered on an outpatient basis. Treatment will be repeated every 28 days. Doxil is administered on day 1 (rate: 1mg/min). Dose levels 1, 2 and 3 (mg/m2 i.v.) are 25, 30 and 30, respectively.
  There is no data to report. Data for this trial was
Arm/Group | Taxotere and Doxil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Taxotere and Doxil
Serious Adverse Events (participants affected / at risk) | 8/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxotere and Doxil (N=39)
Bacterial meningitis (Infections and infestations) | 1 (1)
Fatique (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Bleeding (General disorders) | 2 (2)
Mouth pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No